SleepFlex™ Treatment of Obstructive Sleep Apnea NCT04726514

June 15, 2023

## **Study Protocol (Summary)**

Study participants with mild to moderate obstructive sleep apnea (OSA) underwent 12 weeks of active treatment with the SleepFlex™ program of head and neck exercises.

Statistical analysis includes paired t-tests to evaluate primary and exploratory outcomes in participants who completed the study.

## **Results Summary**

Enrolled participants: 10

Participants with data for analysis: 7

Outcomes are presented as baseline vs. 12-week measures

Total AHI: 15.5±5.1 vs. 12.2±5.5 events/hour (p=0.11)

Supine AHI: 21.0±10.8 vs. 15.3±6.0 events/hour (p=0.048)

Non-supine AHI: 7.3±7.4 vs. 6.8±6.7 events/hour (p=0.064)

Maximal inspiratory pressure: 93±35 vs. 114±34 kPa (p=0.02)

Maximal expiratory pressure: 108±33 vs. 137±14 kPa (p=0.04)

Anterior tongue strength: 53±13 vs. 56±10 kPa (p=0.20)